CLINICAL TRIAL: NCT05292716
Title: Mitral Regurgitation Treatment in Advanced Heart Failure
Acronym: MITRADVANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Marianna Adamo, Principal investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NP4918
Record Dates: First submitted 2022-02-20; First posted 2022-03-23 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Mitral Regurgitation
Keywords: Heart Failure; Mitral Regurgitation; MitraClip; Optimal medical therapy
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MitraClip + Optimal medical therapy (Experimental): Patients randomized to this arm will receive percutaneous treatment of secondary mitral regurgitation by MitraClip system and Optimal medical therapy (OMT) for heart failure
  Interventions: Device: MitraClip
- Optimal medical therapy (No Intervention): Patients randomized to this arm will receive only Optimal medical therapy (OMT) for heart failure

INTERVENTIONS:
Device: MitraClip — MitraClip
  Arms: MitraClip + Optimal medical therapy

SUMMARY:
MITRADVANCE-HF is a prospective, randomized, parallel-controlled, open-label, multicentre study trial enrolling patients with SMR and advanced HF on maximally tolerated standard of care therapies for HF according to the most recent guidelines. Enrolled patients will be randomly assigned, in a 1:1 ratio, to a device arm consisting of MitraClip therapy added to optimal medical therapy (OMT) or a control arm of OMT alone. Approximately 20 Italian high-volume centres will be involved. Enrolment duration will be of 24 months. Follow-up visit will be performed at 3, 6, and 12 months. Primary end-point was the absolute change in overall KCCQ summary score (KCCQ-OS) from baseline to 3 months follow-up.

DETAILED DESCRIPTION:
There are no studies comparing MitraClip and optimal medical therapy (OMT) in patients with advanced heart failure (HF).

The aim of this study is to assess the effects of MitraClip on health status, measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ), in patients with secondary mitral regurgitation (SMR) and advanced HF.

Secondary aims are to evaluate persistence of such benefits up to 1 year as well as changes in survival, HF hospitalization, functional status, symptoms, echocardiographic parameters, and further optimization in medical therapies.

MITRADVANCE-HF is a prospective, randomized, parallel-controlled, open-label, multicenter study trial enrolling patients with SMR and advanced HF on maximally tolerated standard of care therapies for HF according to the most recent guidelines. Enrolled patients will be randomly assigned, in a 1:1 ratio, to a device arm consisting of MitraClip therapy added to optimal medical therapy (OMT) or a control arm of OMT alone. Primary end-point was the absolute change in overall KCCQ summary score (KCCQ-OS) from baseline to 3 months follow-up. A total of 172 patients should be recruited (86 in the device arm and 86 in the control arm. Approximately 20 Italian centers are involved. All screened patients need to be approved by an eligibility committee before randomization. Visit 0 will be performed before randomization. A discharge visit will be performed in patients randomized to the device arm. Visit 1, 2 and 3 will be performed at 3, 6 and 12 months after the randomization in both arms. Transthoracic echocardiography performed during Visit 0, 1, 2 and 3 will be collected and analyzed by an independent Core Laboratory. Adverse events will be adjudicated by an independent committee. Enrolment duration will be of 24 months. The primary completion is the date when the last enrolled subject is assessed for the collection of the primary endpoint. The end of the study is when the last enrolled subject has completed the last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Significant secondary mitral regurgitation (effective regurgitant orifice area ≥ 5 30mm2) confirmed at the end of the screening period
* Optimal medical therapy (OMT) according to recent guidelines.
* Advanced heart failure defined as the presence of all the following criteria, despite OMT:

  * Severe and persistent symptoms of HF (NYHA class III or IV)
  * Severe cardiac dysfunction defined by a reduced left ventricular ejection fraction (LVEF) ≤35% and/or high BNP or NTproBNP levels (BNP>125 pg/ml or NTproBNP>400 pg/ml if sinus rhythm; BNP>375 pg/ml or NTproBNP>1200 pg/ml if atrial fibrillation)
  * Impairment of quality of life (KCCQ < 75 points) AND severe impairment of exercise capacity with inability to exercise or low 6MWT distance (<450 meters) or pVO2 (<14 mL/kg/min or <50% of predicted) OR at least 1 unplanned visit or hospitalization in the last 12 months, due to HF, and requiring intravenous diuretics and/or inotropes.

Exclusion Criteria:

* Unfavorable mitral valve anatomy, which implanting investigator judges as not successfully treatable by the MitraClip (i.e. mitral valve area <3 mm2, leaflet length <7 mm)
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e., noncompliant, perforated)
* Active infections requiring current antibiotic therapy
* Transesophageal echocardiography (TEE) contraindicated or at high risk
* Untreated significant coronary artery disease requiring revascularization
* Iron deficiency defined as serum ferritin <100 μg/L, or ferritin between 100-299 μg/L and transferrin saturation <20% and/or intravenous ferric carboxymaltose administration during the 30 days before randomization
* Coronary artery bypass graft, percutaneous coronary intervention, transcatheter aortic valve replacement or cardiac resynchronization therapy within the prior 30 days
* Pulmonary vein ablation or cardioversion leading to restore of sinus rhythm or AV node ablation in the last 30 days
* Myocardial infarction or cerebrovascular accident within prior 30 days
* Hemodynamic instability defined as systolic blood pressure < 90mmHg and cardiogenic shock or need for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
* Chronic obstructive pulmonary disease, malignancy, or other comorbidities as the main cause of severe symptoms and impaired quality of life.
* Life expectancy <12 months due to non-cardiac conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-04-21 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Absolute change in overall KCCQ summary score (KCCQ-OS) | from baseline to 3 months
  Freedom from all-cause death or unplanned HF events and KCCQ overall summary score (KCCQ-OS) improvement > or =5 points from baseline, at 3 months.

SECONDARY OUTCOMES:
Composite of all-cause death or unplanned HF hospitalization or change in KCCQ-OS | from baseline to 3, 6 and 12 months
  Unplanned HF hospitalization is defined as Admission to an inpatient unit or ward in the hospital for ≥24 h, including an emergency department stay with symptoms, signs and/or laboratory evidence of worsening heart failure; pulmonary edema, administration of intravenous therapies (loop diuretic agents, vasodilators, inotropic agents, vasopressors) or mechanical heart failure therapies (ultrafiltration, cardiac resynchronization, IABP, LVAD); hospitalizations requiring oxygen therapy.
  Kansas City Cardiomyopathy Questionnaire (KCCQ) aims at evaluating quality of life in heart failure patients using a scale including 100 points (from 0 [worst] to 100 [best]).
All-cause death | at 3 months, 6 and 12 months
Cardiovascular death | at 3 months, 6 and 12 months
  Defined according to MVARC-2 definition as death due to Heart Failure, Myocardial Infarction, Major/Disabling Bleeding, Thromboembolism, Stroke, Arrythmia, Cardiovascular Infection, Cardiac Tamponade, Sudden Death, Device Failure
Unplanned HF hospitalization | at 3, 6 and 12 months
  Admission to an inpatient unit or ward in the hospital for ≥24 h, including an emergency department stay with symptoms, signs and/or laboratory evidence of worsening heart failure; pulmonary edema, administration of intravenous therapies (loop diuretic agents, vasodilators, inotropic agents, vasopressors) or mechanical heart failure therapies (ultrafiltration, cardiac resynchronization, IABP, LVAD); hospitalizations requiring oxygen therapy.
Absolute change in KCCQ-OS | from baseline to 6 and 12 months
  Kansas City Cardiomyopathy Questionnaire aims at evaluating quality of life in heart failure patients using a scale including 100 points (from 0 [worst] to 100 [best])
Recurrent HF events | at 3, 6 and 12 months

OTHER OUTCOMES:
Absolute change in EQ-5D | from baseline to 3, 6 and 12 months
  The EQ-5D questionnaire is standardized instrument for measuring generic health status using five dimensions. Each dimension has 5 levels. The final number is included between 0 and 1 (0=worst and 1=best)
Patients' Global Impression of Change (PGIC) Scale | at 3, 6 and 12 months
  The Patients' Global Impression of Change (PGIC) Scale will assess the degree of change in patient's health status in terms of overall improvement (very much improved, much improved, minimally improved, unchanged, minimally worse, much worse, very much worse.
Change in NYHA class | from baseline to 3, 6 and 12 months
  The New York Heart Association scale include 4 level of heart failure symptoms: 1=No limitation of physical activity, ordinary physical activity does not cause undue fatigue or dyspnea; 2= Slight limitation of physical activity, ordinary physical activity results in fatigue or dyspnea; 3: Marked limitation of physical activity, less than ordinary activity causes fatigue or dyspnea; 4=Symptoms of heart failure at rest
Absolute and percentage change in 6-minute walk test (6MWT) distance in meters | from baseline to 3, 6 and 12 months
Absolute change and percentage in NT-proBNP levels in pg/mL | from baseline to 3, 6 and 12 months.
Absolute and percentage change in systolic pulmonary pressure (mmHg) assessed by echocardiography | from baseline to 3, 6 and 12 months
Absolute and percentage change in left atrial volume (mL) | from baseline to 3, 6 and 12 months.
Absolute and percentage change in left ventricular end-diastolic and end-systolic volumes (mL) | from baseline to 3, 6 and 12 months
Absolute and percentage change in right ventricular fractional area change (FAC) (percent) | from baseline to 3, 6 and 12 months
Absolute and percentage change in diuretic dose | from baseline to 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marianna Adamo, Brescia, Lombardy, Italy